CLINICAL TRIAL: NCT04507269
Title: A Phase 2 Randomized, Placebo-Controlled Study in Mainland China to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of VIR-2218
Brief Title: Study of VIR-2218 in Patients With Chronic Hepatitis B in Mainland China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brii Biosciences Limited (Industry)
Collaborators: Vir Biotechnology, Inc. (Industry); Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIR-2218-1005
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B Virus; Chronic Hepatitis B; HBV; Hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- VIR-2218 (Experimental): Drug: VIR-2218 VIR-2218 given by subcutaneous injection
  Interventions: Drug: VIR-2218
- Placebo (Placebo Comparator): Drug: Placebo Saline given by subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIR-2218 — VIR-2218 given by subcutaneous injection
  Arms: VIR-2218
Drug: Placebo — Saline given by subcutaneous injection
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety, pharmacokinetics characteristics, and antiviral activities of multiple doses of VIR-2218 in adults with chronic HBV infection in mainland China.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 - 65;
* Weight ≥ 40 kg to ≤ 125 kg;
* Chronic HBV infection as defined by a positive serum HBsAg for ≥ 6 months;

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation;
* Significant fibrosis or cirrhosis;
* History or evidence of drug or alcohol abuse;
* History of intolerance to SC injection;
* History of chronic liver disease from any cause other than chronic HBV infection;
* History of hepatic decompensation;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Chen, Study Director — Brii Biosciences Limited
Locations (2):
- China (2):
  - Investigative Site, Beijing, Beijing Municipality
  - Investigative Site, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: VIR-2218 50 mg: HBeAg negative, participants received 2 SC doses of VIR-2218 50 mg administered 4 weeks apart
- Part 1: VIR-2218 100 mg: HBeAg negative, participants received 2 SC doses of VIR-2218 100 mg administered 4 weeks apart
- Part 1: Placebo: HBeAg negative, participants received 2 SC doses of placebo administered 4 weeks apart
- Part 2: VIR-2218 50mg: HBeAg positive, participants received 2 SC doses of VIR-2218 50 mg administered 4 weeks apart
- Part 2: VIR-2218 100 mg: HBeAg positive, participants received 2 SC doses of VIR-2218 100 mg administered 4 weeks apart
- Part 2: Placebo: HBeAg positive, participants received 2 SC doses of placebo administered 4 weeks apart
Period: Overall Study
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 1: Placebo | Part 2: VIR-2218 50mg | Part 2: VIR-2218 100 mg | Part 2: Placebo
Started | 4 | 4 | 3 | 4 | 4 | 2
Dosed | 4 | 4 | 3 | 4 | 4 | 2
Completed | 3 | 3 | 3 | 4 | 3 | 2
Not Completed | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: VIR-2218 50 mg: HBeAg negative, participants received 2 SC doses of VIR-2218 50 mg administered every 4 weeks apart
- Part 1: VIR-2218 100 mg: HBeAg negative, participants received 2 SC doses of VIR-2218 100 mg administered every 4 weeks apart
- Part 1: Placebo: HBeAg negative, participants received 2 SC doses of placebo administered every 4 weeks apart
- Part 2: VIR-2218 50 mg: HBeAg positive, participants received 2 SC doses of VIR-2218 50 mg administered every 4 weeks apart
- Part 2: VIR-2218 100 mg: HBeAg positive, participants received 2 SC doses of VIR-2218 100 mg administered every 4 weeks apart
- Part 2: Placebo: HBeAg positive, participants received 2 SC doses of placebo administered every 4 weeks apart
- Total: Total of all reporting groups
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 1: Placebo | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg | Part 2: Placebo | Total
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 4 | 2 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (9.68) | 36.5 (9.26) | 31.0 (5.20) | 41.8 (4.27) | 39.5 (10.66) | 38.0 (11.31) | 39.7 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Male | 4 | 4 | 3 | 3 | 3 | 1 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 4 | 3 | 4 | 4 | 2 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 4 | 4 | 3 | 4 | 4 | 2 | 21
Baseline log10 hepatitis B surface antigen [Mean (Standard Deviation); unit: log10 IU/mL] | 2.815 (0.4865) | 3.278 (0.7910) | 2.948 (0.4822) | 3.598 (0.5479) | 3.243 (0.4848) | 3.722 (0.0729) | 3.239 (0.5756)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with treatment-emergent adverse events (TEAEs) as assessed by CTCAE v5.0 are summarized by cohort. Incidence is defined as the number of participants with TEAEs in relation to the total number of participants in the cohort. TEAEs are defined as any AEs with an onset date of on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug.
Time Frame: up to 48 weeks
Population: All randomized participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 1: Placebo | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg | Part 2: Placebo
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 4 | 2
Participants
  Any TEAEs | 1 | 2 | 0 | 2 | 1 | 1
  Any TEAEs of CTCAE Grade 1 | 0 | 1 | 0 | 2 | 1 | 1
  Any TEAEs of CTCAE Grade 2 | 1 | 1 | 0 | 0 | 0 | 0
  Any TEAEs of CTCAE Grade 3 or above | 0 | 0 | 0 | 0 | 0 | 0
  Any drug related TEAEs | 0 | 0 | 0 | 1 | 1 | 0
  Any serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Clinical Assessments Including But Not Limited to Laboratory Test Results
Description: Number of participants with graded hematology, coagulation, chemistry abnormalities, and clinically significant abnormalities in vital signs and ECGs
Time Frame: up to 48 weeks
Population: All randomized participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 1: Placebo | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg | Part 2: Placebo
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 4 | 2
Participants
  Any post baseline laboratory abnormalities of CTCAE Grade 1 | 4 | 4 | 2 | 2 | 4 | 2
  Any post baseline laboratory abnormalities of CTCAE Grade 2 or above | 0 | 0 | 0 | 0 | 0 | 0
  Any clinically significant vital signs | 0 | 0 | 0 | 0 | 0 | 0
  Any clinically significant ECGs | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: PK: Maximum Plasma Concentration
Description: VIR-2218 and metabolite maximum plasma concentrations (ng/mL)
  VIR-2218 and metabolite concentrations were tested at predose on Day 1 and 1h, 2h, 4h, 8h, and 24h postdose, Week 1, predose on Week 4 and 1h, 2h, 4h, 8h, and 24h postdose, Week 5, Week 8, Week 16, and Week 24.
Time Frame: Maximum plasma concentrations were calculated based on all above results for Day 1 and Day 29 (Week 4).
Population: All randomized participants who received at least 1 dose of VIR-2218 and had 1 post-baseline PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2: VIR-2218 50 mg: HBeAg positive, participants received 2 SC doses of VIR-2218 50 mg administered 4 weeks apart
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng/mL
  VIR-2218 Cmax (Day 1): number analyzed (Participants) | 4 | 4 | 3 | 3
  VIR-2218 Cmax (Day 1) | 120 (40.5) | 144 (100.5) | 65.8 (58.6) | 260 (90.4)
  VIR-2218 Cmax (Day 29): number analyzed (Participants) | 2 | 4 | 4 | 4
  VIR-2218 Cmax (Day 29) | 125 (48.8) | 198 (52.9) | 76.5 (35.7) | 268 (43.0)
  AS(N-1)3'VIR-2218 Cmax (Day 1): number analyzed (Participants) | 1 | 1 | 0 | 2
  AS(N-1)3'VIR-2218 Cmax (Day 1) | 10.2 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 31.4 (NA) — %Geometric CoV not reported; measurable in 1/4 participants |  | 28.1 (171.1)
  AS(N-1)3'VIR-2218 Cmax (Day 29): number analyzed (Participants) | 1 | 2 | 2 | 2
  AS(N-1)3'VIR-2218 Cmax (Day 29) | 16.3 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 23.6 (48.8) | 9.75 (1.1) | 19.3 (82.1)

4. Secondary Outcome: PK: Time to Reach Maximum Plasma Concentration
Description: VIR-2218 and metabolite time to Cmax (h)
  VIR-2218 and metabolite concentrations were tested at predose on Day 1 and 1h, 2h, 4h, 8h, and 24h postdose, Week 1, predose on Week 4 and 1h, 2h, 4h, 8h, and 24h postdose, Week 5, Week 8, Week 16, and Week 24.
Time Frame: Time to Cmax were calculated based on all above results for Day 1 and Day 29 (Week 4).
Population: All randomized participants who received at least 1 dose of VIR-2218 and had 1 post-baseline PK parameter
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
hour
  VIR-2218 Tmax (Day 1) | 4.99 [1.88 to 8.03] | 2.00 [0.967 to 8.08] | 4.02 [4.00 to 7.80] | 4.00 [4.00 to 7.58]
  VIR-2218 Tmax (Day 29) | 7.76 [1.08 to 8.13] | 4.02 [2.00 to 7.85] | 2.50 [0.967 to 4.00] | 5.93 [1.00 to 8.02]
  AS(N-1)3'VIR-2218 Tmax (Day 1): number analyzed (Participants) | 3 | 2 | 2 | 4
  AS(N-1)3'VIR-2218 Tmax (Day 1) | 7.95 [3.98 to 8.05] | 4.98 [2.03 to 7.92] | 7.80 [7.80 to 7.80] | 5.79 [4.00 to 22.1]
  AS(N-1)3'VIR-2218 Tmax (Day 29): number analyzed (Participants) | 4 | 4 | 2 | 4
  AS(N-1)3'VIR-2218 Tmax (Day 29) | 7.76 [4.05 to 8.13] | 5.93 [2.00 to 8.03] | 4.00 [4.00 to 4.00] | 5.93 [4.00 to 8.02]

5. Secondary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve to Last Measurable Timepoint
Description: VIR-2218 and metabolite area under the curve from time 0 to last measurable time (ng*h/mL)
  VIR-2218 and metabolite concentrations were tested at predose on Day 1 and 1h, 2h, 4h, 8h, and 24h postdose, Week 1, predose on Week 4 and 1h, 2h, 4h, 8h, and 24h postdose, Week 5, Week 8, Week 16, and Week 24.
Time Frame: Area under the curve were calculated based on all above results for Day 1 and Day 29 (Week 4).
Population: All randomized participants who received at least 1 dose of VIR-2218 and had 1 post-baseline PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng*h/mL
  VIR-2218 AUClast (Day 1) | 1080 (25.3) | 1400 (115.6) | 626 (31.1) | 3190 (42.3)
  VIR-2218 AUClast (Day 29) | 854 (34.2) | 2390 (26.6) | 580 (56.9) | 3140 (15.8)
  AS(N-1)3'VIR-2218 AUClast (Day 1): number analyzed (Participants) | 3 | 2 | 2 | 4
  AS(N-1)3'VIR-2218 AUClast (Day 1) | 58.7 (28.9) | 159 (30.5) | 67.6 (2.1) | 180 (63.4)
  AS(N-1)3'VIR-2218 AUClast (Day 29): number analyzed (Participants) | 4 | 4 | 2 | 4
  AS(N-1)3'VIR-2218 AUClast (Day 29) | 50.2 (52.5) | 140 (81.2) | 63.1 (6.1) | 155 (39.8)

6. Secondary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve to Infinity
Description: VIR-2218 and metabolite area under the curve from time 0 to infinity (ng*h/mL)
  VIR-2218 and metabolite concentrations were tested at predose on Day 1 and 1h, 2h, 4h, 8h, and 24h postdose, Week 1, predose on Week 4 and 1h, 2h, 4h, 8h, and 24h postdose, Week 5, Week 8, Week 16, and Week 24.
Time Frame: Area under the curve were calculated based on all above results for Day 1 and Day 29 (Week 4).
Population: All randomized participants who received at least 1 dose of VIR-2218 and had 1 post-baseline PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng*h/mL
  VIR-2218 AUCinf (Day 1): number analyzed (Participants) | 0 | 2 | 0 | 0
  VIR-2218 AUCinf (Day 1) |  | 2820 (16.7) |  |
  VIR-2218 AUCinf (Day 29): number analyzed (Participants) | 0 | 1 | 1 | 1
  VIR-2218 AUCinf (Day 29) |  | 2570 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 1210 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 3530 (NA) — %Geometric CoV not reported; measurable in 1/4 participants
  AS(N-1)3'VIR-2218 AUCinf (Day 1): number analyzed (Participants) | 0 | 0 | 0 | 0
  AS(N-1)3'VIR-2218 AUCinf (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: PK: Percent of Area Extrapolated From AUC Last to Infinity
Description: VIR-2218 and metabolite percent of area extrapolated from AUC last to infinity (%)
  VIR-2218 and metabolite concentrations were tested at predose on Day 1 and 1h, 2h, 4h, 8h, and 24h postdose, Week 1, predose on Week 4 and 1h, 2h, 4h, 8h, and 24h postdose, Week 5, Week 8, Week 16, and Week 24.
Time Frame: Percent of area extrapolated from AUC last to infinity were calculated based on all above results for Day 1 and Day 29 (Week 4).
Population: All randomized participants who received at least 1 dose of VIR-2218 and had 1 post-baseline PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % of AUCinf
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
% of AUCinf
  VIR-2218 %AUCextrap (Day 1): number analyzed (Participants) | 0 | 2 | 0 | 0
  VIR-2218 %AUCextrap (Day 1) |  | 2.69 (5.1) |  |
  VIR-2218 %AUCextrap (Day 29): number analyzed (Participants) | 1 | 1 | 2 | 1
  VIR-2218 %AUCextrap (Day 29) | 46.2 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 13.8 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 23.9 (263.4) | 5.88 (NA) — %Geometric CoV not reported; measurable in 1/4 participants
  AS(N-1)3'VIR-2218 %AUCextrap (Day 1): number analyzed (Participants) | 0 | 0 | 0 | 0
  AS(N-1)3'VIR-2218 %AUCextrap (Day 29): number analyzed (Participants) | 0 | 1 | 0 | 0
  AS(N-1)3'VIR-2218 %AUCextrap (Day 29) |  | 49.2 (NA) — %Geometric CoV not reported; measurable in 1/4 participants |  |

8. Secondary Outcome: PK: Apparent Terminal Elimination Half-life
Description: VIR-2218 and metabolite apparent terminal elimination half-life (h)
  VIR-2218 and metabolite concentrations were tested at predose on Day 1 and 1h, 2h, 4h, 8h, and 24h postdose, Week 1, predose on Week 4 and 1h, 2h, 4h, 8h, and 24h postdose, Week 5, Week 8, Week 16, and Week 24.
Time Frame: Apparent terminal elimination half-life were calculated based on all above results for Day 1 and Day 29 (Week 4).
Population: All randomized participants who received at least 1 dose of VIR-2218 and had 1 post-baseline PK parameter
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
hour
  VIR-2218 t1/2 (Day 1): number analyzed (Participants) | 0 | 2 | 0 | 0
  VIR-2218 t1/2 (Day 1) |  | 4.16 [4.10 to 4.22] |  |
  VIR-2218 t1/2 (Day 29): number analyzed (Participants) | 0 | 1 | 1 | 1
  VIR-2218 t1/2 (Day 29) |  | 7.66 [7.66 to 7.66] | 6.53 [6.53 to 6.53] | 5.49 [5.49 to 5.49]
  AS(N-1)3'VIR-2218 t1/2 (Day 1): number analyzed (Participants) | 0 | 0 | 0 | 0
  AS(N-1)3'VIR-2218 t1/2 (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: PK: Apparent Plasma Clearance
Description: VIR-2218 and metabolite apparent plasma clearance CL/F (mL/h)
  VIR-2218 and metabolite concentrations were tested at predose on Day 1 and 1h, 2h, 4h, 8h, and 24h postdose, Week 1, predose on Week 4 and 1h, 2h, 4h, 8h, and 24h postdose, Week 5, Week 8, Week 16, and Week 24.
Time Frame: Apparent plasma clearance were calculated based on all above results for Day 1 and Day 29 (Week 4).
Population: All randomized participants who received at least 1 dose of VIR-2218 and had 1 post-baseline PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
mL/h
  VIR-2218 CL/F (Day 1): number analyzed (Participants) | 0 | 2 | 0 | 0
  VIR-2218 CL/F (Day 1) |  | 35400 (16.7) |  |
  VIR-2218 CL/F (Day 29): number analyzed (Participants) | 0 | 1 | 1 | 1
  VIR-2218 CL/F (Day 29) |  | 39000 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 41300 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 28300 (NA) — %Geometric CoV not reported; measurable in 1/4 participants
  AS(N-1)3'VIR-2218 CL/F (Day 1): number analyzed (Participants) | 0 | 0 | 0 | 0
  AS(N-1)3'VIR-2218 CL/F (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: PK: Apparent Volume of Distribution
Description: VIR-2218 and metabolite apparent volume of distribution Vz/F (mL)
  VIR-2218 and metabolite concentrations were tested at predose on Day 1 and 1h, 2h, 4h, 8h, and 24h postdose, Week 1, predose on Week 4 and 1h, 2h, 4h, 8h, and 24h postdose, Week 5, Week 8, Week 16, and Week 24.
Time Frame: Apparent volume of distribution were calculated based on all above results for Day 1 and Day 29 (Week 4).
Population: All randomized participants who received at least 1 dose of VIR-2218 and had 1 post-baseline PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
mL
  VIR-2218 Vz/F (Day 1): number analyzed (Participants) | 0 | 2 | 0 | 0
  VIR-2218 Vz/F (Day 1) |  | 213000 (18.6) |  |
  VIR-2218 Vz/F (Day 29): number analyzed (Participants) | 0 | 1 | 1 | 1
  VIR-2218 Vz/F (Day 29) |  | 431000 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 389000 (NA) — %Geometric CoV not reported; measurable in 1/4 participants | 224000 (NA) — %Geometric CoV not reported; measurable in 1/4 participants
  AS(N-1)3'VIR-2218 Vz/F (Day 1): number analyzed (Participants) | 0 | 0 | 0 | 0
  AS(N-1)3'VIR-2218 Vz/F (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Maximum Change of Serum HBsAg From Baseline
Description: Maximum change of serum HBsAg from Day 1 until 12 weeks post last dose (negative values mean reductions from baseline, positive values mean increased from baseline)
Time Frame: up to 16 weeks
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 non-missing data for antiviral parameters
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 1: Placebo | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg | Part 2: Placebo
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 4 | 2
log10 IU/mL | -1.064 (0.1047) | -1.346 (0.5169) | -0.049 (0.0158) | -0.793 (0.1017) | -1.268 (0.1693) | -0.120 (0.0826)

12. Secondary Outcome: Number of Participants With Serum HBsAg Loss
Description: Number of participants with serum HBsAg < 0.05 IU/mL at two or more consecutive measurements
Time Frame: up to 48 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 1: Placebo | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg | Part 2: Placebo
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 4 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Sustained Serum HBsAg Loss for at Least 6 Months
Description: Number of participants with sustained serum HBsAg < 0.05 IU/mL at all visits for at least 6 months
Time Frame: up to 48 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 1: Placebo | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg | Part 2: Placebo
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 4 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Anti-HBs Seroconversion at Any Timepoint
Description: Anti-HBs seroconversion is defined as anti-HBs positivity at two or more consecutive measurements
Time Frame: up to 48 weeks
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 non-missing data for antiviral activity parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg | Part 1: Placebo | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg | Part 2: Placebo
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 4 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 0

15. Secondary Outcome: For HBeAg-positive Subjects: Number of Subjects With HBeAg Loss and/or Anti-HBe Seroconversion at Any Timepoint
Description: HBeAg loss is defined as quantitative HBeAg < 0.14 IU/mL at two or more consecutive measurements. Anti-HBe seroconversion is defined as anti-HBe positivity at two or more consecutive measurements.
Time Frame: up to 48 weeks
Population: Part 2 (HBeAg positive) participants only; all randomized participants who received at least 1 dose of study drug and had at least 1 non-missing data for antiviral activity parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg | Part 2: Placebo
Number analyzed (Participants) | 4 | 4 | 2
Participants
  HBeAg loss | 0 | 0 | 0
  Anti-HBe seroconversion | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 48 weeks after the first dose of VIR-2218 or placebo
Groups:
- Part 1: VIR-2218 100 mg 100 mg: HBeAg negative, participants received 2 SC doses of VIR-2218 100 mg administered every 4 weeks apart
Arm/Group | Part 1: VIR-2218 50 mg | Part 1: VIR-2218 100 mg 100 mg | Part 1: Placebo | Part 2: VIR-2218 50 mg | Part 2: VIR-2218 100 mg | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/3 | 0/4 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3 | 0/4 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 1/4 | 2/4 | 0/3 | 2/4 | 1/4 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: VIR-2218 50 mg (N=4) | Part 1: VIR-2218 100 mg 100 mg (N=4) | Part 1: Placebo (N=3) | Part 2: VIR-2218 50 mg (N=4) | Part 2: VIR-2218 100 mg (N=4) | Part 2: Placebo (N=2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will submit the proposed publication to sponsor at least 60 days prior to submission to a publisher.

Sponsor shall advise investigator any information that are confidential or may impair the availability of patent protection for study inventions.

Sponsor may require to remove confidential information and/or to delay the proposed publication or presentation for an additional 60 days to seek patent protection for study inventions.

DOCUMENTS (2):
  • Study Protocol (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT04507269/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT04507269/SAP_001.pdf